CLINICAL TRIAL: NCT01050283
Title: A Multicenter Trial to Evaluate 18F-FDG Uptake by PET in Patients With Advanced Pancreatic Adenocarcinoma as an Early Indicator of Drug Activity
Brief Title: A Study to Evaluate [18F]-FDG PET (Fluorodeoxyglucose-positron) in Patients With Pancreatic Cancer (MK-0000-144)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-144; 144
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Advanced Pancreatic Adenocarcinoma
Keywords: Advanced pancreatic adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): [18F]-FDG-PET/CT (Computed Tomography) Imaging
  Interventions: Procedure: Comparator: [18F]-FDG PET/CT and Volumetric CT

INTERVENTIONS:
Procedure: Comparator: [18F]-FDG PET/CT and Volumetric CT — Patients will receive gemcitabine-based therapy as prescribed by their treating physician. FDG-PET/CT scans will be performed at baseline following enrollment, and after 3 and 6-7 weeks of therapy. Volumetric CT scans will be performed at baseline following enrollment, and after 3 and 6-7 weeks of therapy.

SUMMARY:
This study will determine whether [18F]-fluorodeoxyglucose-positron emission tomography (FDG-PET) can be used to screen for the activity of novel pancreatic cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of Stage IV pancreatic adenocarcinoma with distant metastases
* Patient is scheduled to receive standard chemotherapy containing gemcitabine
* Patient has not received prior systemic therapy for advanced pancreatic adenocarcinoma
* Patient must be available for periodic blood sampling, study-related assessments, and management at the treating institution

Exclusion Criteria:

* Patient has had open abdominal surgery within 6 weeks of the screening visit
* Patient has had radiotherapy to the thorax, abdomen, or pelvis within 6 months of the screening visit
* Patient has an active infection, inflammation, or unresolved bowel obstruction
* Patient has poorly controlled diabetes

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Association of changes in FDG uptake with overall survival (OS) | Week 3 and at least 7 months after the last patient is treated

SECONDARY OUTCOMES:
Association of metabolic response with OS | Baseline, Week 3, and at least 7 months after the last patient is treated
Correlation between FDG standardized uptake values (SUV) at Week 3 and Week 6-7 | Week 3 and Week 6-7

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC